CLINICAL TRIAL: NCT03191643
Title: 18F-FDG PET-guided External Beam Radiotherapy in Iodine-refractory Differentiated Thyroid Cancer
Brief Title: PET-guided External Beam Radiotherapy in Differentiated Thyroid Cancer
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Alessio Giuseppe Morganti, Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: Thyroid-COBRA
Record Dates: First submitted 2017-06-15; First posted 2017-06-19 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Differentiated Thyroid Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- differentiated thyroid cancer: Patients with locally recurrent thyroid cancer, treated with radical radiotherapy after total thyroidectomy +/- central compartment and/or laterocervical lymphadenectomy, previously treated with one or more cycles of 131 Iodine-ablation (RAI) and TSH suppression.

SUMMARY:
Description of the role of a post-operative external beam radiotherapy in patients with differentiated thyroid cancer.

DETAILED DESCRIPTION:
The role of post-operative external beam radiotherapy (EBRT) in differentiated thyroid cancer is still discussed considering the low clinical aggressiveness and the availability of ablative 131Iodine therapy. However, there is a subgroup of tumors which lose the ability to capture Iodine over time. This study wants to describe the role of a post-operative external beam radiotherapy in patients with differentiated thyroid cancer.

ELIGIBILITY:
Inclusion Criteria:

* detectable thyroglobulin (Tg),
* negative post-metabolic radiotherapy whole body scintigraphy,
* no surgical indications.

Exclusion Criteria:

* prior radiotherapy in the head and neck area
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally recurrent thyroid cancer, treated with radical external beam radiotherapy (EBRT) after total thyroidectomy +/- central compartment and/or laterocervical lymphadenectomy, previously treated with one or more cycles of 131 Iodine-ablation (RAI) and TSH suppression.
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2011-10-01 (Actual); Primary Completion 2016-01-31 (Actual); Study Completion 2016-01-31 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 6 months
  Progression-free survival (PFS) after radiotherapy is evaluated with CT-scan and 18F FDG PET-scan. Also laboratory tests are performed (HTG serum level evaluation in case of biochemical recurrence).

SECONDARY OUTCOMES:
toxicities | 6 months
  Acute and late toxicities after radiotherapy are assessed with CTCAE v. 4.03 and EORTC-RTOG scales, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Alessio G. Morganti, MD, Study Director — Radiation Oncology Center, Department of Experimental, Diagnostic and Specialty Medicine - DIMES, University of Bologna, S.Orsola-Malpighi Hospital, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Farina E, Monari F, Castellucci P, Romani F, Repaci A, Farina A, Zanirato Rambaldi G, Frezza G, Mazzarotto R, Cammelli S, Tagliaferri L, Autorino R, Deodato F, Macchia G, Cilla S, Valentini V, Fanti S, Morganti AG. 18F-FDG Pet-Guided External Beam Radiotherapy in Iodine-Refractory Differentiated Thyroid Cancer: A Pilot Study. J Thyroid Res. 2017;2017:9807543. doi: 10.1155/2017/9807543. Epub 2017 Oct 19. PMID 29201490